CLINICAL TRIAL: NCT06470932
Title: Outcome of Patients Admitted to Pediatric Intensive Care for Acute Respiratory Failure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, EssaiClinique_SUIVIRA, Clinical professor, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC23.0449
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Respiratory Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow up (Experimental)
  Interventions: Diagnostic Test: Follow-up consult

INTERVENTIONS:
Diagnostic Test: Follow-up consult — Patients will be ask to participate to a follow-up consult

SUMMARY:
This study aims to assess the quality of life of patients six months after admission to a pediatric intensive care unit for acute respiratory failure. Children's quality of life will be assessed using the PedsQL scale at 6 months. This is a prospective cohort diagnostic and prognostic study.

ELIGIBILITY:
Inclusion Criteria:

* admitted in the PICU of Grenoble-Alps University Hospital
* for acute respiratory failure (code J960) requiring mechanical ventilation for at least 48hrs

Exclusion Criteria:

* already followed-up by a pediatric pulmonologist
* with congenital disease
* with long term ventilation
* still admitted at 3 months

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Quality of life at 3 months | 3 months
  Quality of life at 3 months measured by PEDS QL (Pediatric Quality of Life) scale, scoring from 0 (good quality of life) to 92 (poor quality of life)

IPD SHARING:
Plan to Share IPD: No